CLINICAL TRIAL: NCT00336063
Title: A Phase I Trial of 5Azacitidine and Suberoylanilide Hydroxamic Acid in Patients With Metastatic or Locally Recurrent Nasopharyngeal Carcinoma and Nasal NK-T Cell Lymphoma
Brief Title: Vorinostat and Azacitidine in Treating Patients With Locally Recurrent or Metastatic Nasopharyngeal Cancer or Nasal Natural Killer T-Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00089; NCI-2009-00089 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-6837; CTRG NP03/19/04; CDR0000472702; CTRG NP03/19/04 (Other: Johns Hopkins Singapore); 6837 (Other: CTEP); P30CA006973 (NIH)
Record Dates: First submitted 2006-06-08; First posted 2006-06-12 (Estimated); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Adult Nasal Type Extranodal NK/T-Cell Lymphoma; Recurrent Nasopharyngeal Keratinizing Squamous Cell Carcinoma; Recurrent Nasopharyngeal Undifferentiated Carcinoma; Stage IV Nasopharyngeal Keratinizing Squamous Cell Carcinoma AJCC v7; Stage IV Nasopharyngeal Undifferentiated Carcinoma AJCC v7
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — Azacitidine; Vorinostat

ARMS (1):
- Treatment (azacitidine, vorinostat) (Experimental): Patients receive azacitidine SC on days 1-10 and vorinostat PO BID on days 1-14. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Vorinostat

INTERVENTIONS:
Drug: Azacitidine — Given SC
  Other Names: 5 AZC; 5-AC; 5-Azacitidine; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Vorinostat — Given PO
  Other Names: L-001079038; MSK-390; SAHA; Suberanilohydroxamic Acid; Suberoylanilide Hydroxamic Acid; Zolinza

SUMMARY:
This phase I trial studies the side effects and best dose of vorinostat when given together with azacitidine in treating patients with nasopharyngeal cancer or nasal natural killer T-cell lymphoma that has recurred (come back) at or near the same place as the original (primary) tumor, usually after a period of time during which the cancer could not be detected or has spread to other parts of the body. Drugs used in chemotherapy, such as vorinostat and azacitidine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Vorinostat and azacitidine also may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving vorinostat together with azacitidine may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Define toxicity profile of escalating doses of suberoylanilide hydroxamic acid (SAHA) given in conjunction with a fixed dose of 5 Azacytidine (5AC) (azacitidine) in patients with locally recurrent and metastatic nasopharyngeal carcinoma and natural killer (NK)-T cell nasal lymphoma.

II. Define the biologically optimal dose of SAHA given in conjunction with a fixed dose of 5AC in patients with locally recurrent and metastatic nasopharyngeal carcinoma and NKT cell nasal lymphoma based on evidence of Epstein-Barr virus (EBV) lytic induction in tumor biopsies and plasma.

III. Study the effect of 5AC on the pharmacokinetic of SAHA in patients with locally recurrent and metastatic nasopharyngeal carcinoma and NK-T cell nasal lymphoma.

IV. Assess the effect of SAHA on histone acetylation as measured in tumor and peripheral blood mononuclear cells of patients with locally recurrent and metastatic nasopharyngeal carcinoma and NK-T cell nasal lymphoma V. Assess the effect of 5AC on EBV promoter demethylation as measured in tumor patients with locally recurrent and metastatic nasopharyngeal carcinoma and NK-T cell nasal lymphoma.

OUTLINE: This is a dose-escalation study of vorinostat (SAHA).

Patients receive azacitidine subcutaneously (SC) on days 1-10 and vorinostat orally (PO) twice daily (BID) on days 1-14. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity.

Patients with responding disease may continue treatment at the discretion of the principal investigator. Cohorts of 3-6 patients receive escalating doses of SAHA until the maximum tolerated dose (MTD) is determined.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven nasopharyngeal carcinoma (World Health Organization [WHO] type 3) or extranodal NK-T-cell non-Hodgkin's lymphoma, nasal type (recurrence or metastases does not require tissue documentation)
* Patients must have metastatic disease or locally recurrent disease that is not amendable to surgical resection
* Patients must have locally recurrent disease that is not amendable to further treatment with radiotherapy with curative intent
* Patients must have metastatic disease or locally recurrent disease that has been treated with at least one regimen of chemotherapeutic agents after relapse; patient must be at least 4 weeks since prior chemotherapy or radiation therapy
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy greater than 6 months
* Leukocytes >= 3,000/ul
* Absolute neutrophil count >= 1,500/ul
* Platelets >= 100,000/ul
* Total bilirubin =< 1.5 X normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normal
* Prothrombin time =< 1.5 X normal institutional limits
* Serum albumin >= 2.7 grams/deciliter
* Creatinine =< 1.5 X normal institutional limits or a calculated creatinine clearance of > 50 mls/min
* Sexually active women of child-bearing potential should have a negative serum or urine pregnancy test within 21 days of enrolling on trial; women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Patients must be informed of the investigational nature of the treatment, results that might be expected, and potential toxicities; they must be able to give informed written consent according to federal and institutional guidelines

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents
* Patients with known central nervous system (CNS) involvement (brain metastases or carcinomatous meningitis should be excluded from this clinical trial; patients with skull base involvement are eligible for this study
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to 5AC or SAHA
* Patients should not have taken sodium valproate for at least 2 weeks prior to enrollment
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with 5AC and SAHA
* Human immunodeficiency virus (HIV)-positive patients receiving combination anti-retroviral therapy are excluded from the study
* Patients with chronic active hepatitis B are excluded from the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-03-03 (Actual); Primary Completion 2013-04-19 (Actual); Study Completion 2026-03-19 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of vorinostat and azacitidine, defined as the dose at which less than one-third of patients experience a dose limiting toxicity (i.e., fewer than 2 of 6 patients) | Day 28
  Graded according to the National Cancer Institute/Division of Cancer Treatment Common Toxicity Criteria.
Precision of the estimated dose-response curve based on induction of lytically replicated viral particles in the plasma following treatment | Up to 16 weeks
  A non-parametric and a parametric approach will be used. The non-parametric approach will entail averaging the biologic effects from the patients at each time point, plotting them versus dose, and connecting the points to get the dose-response curve. The parametric approach will use a polynomial regression model with two degrees of freedom for modeling dose. A spline model may also be used.

SECONDARY OUTCOMES:
Pharmacokinetics of vorinostat in patients with locally recurrent and metastatic nasopharyngeal carcinoma and NK-T cell nasal lymphoma | 0, 15, 45, 60, 120, 180, 270, 360, and 480 minutes on days 1 and 14 of course 1
  Performed using a validated high performance liquid chromatography method. Maximum concentration (Cmax) and time to Cmax will be read off the curve, terminal T1/2 will be derived using the slope of the terminal portion of the semilogarithmic concentration-time plot, incorporating at least 3 time points in the extrapolation of the curve. Area-under-the curve (AUC) (infinity) of the semilog plot will be estimated using the trapezoidal method, and oral clearance (CL/F) will be derived using Dose/AUC, volume of distribution will be calculated.
Proportions of patients with high and low histone acetylation | Baseline
  The proportion of patients whose histone acetylation status changes in each group will be estimated with its 95% confidence interval. Percent agreement and kappa will be used.
EBV promoter demethylation as measured in tumor patients with locally recurrent and metastatic nasopharyngeal carcinoma and NK-T cell nasal lymphoma | Baseline
  The proportion of patients whose EBV promoter demethylation status changes in each group will be estimated with its 95% confidence interval. Percent agreement and kappa will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Son Hsieh, Principal Investigator — Johns Hopkins Singapore
Locations (5):
- Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland, United States
- Chinese University of Hong Kong-Prince of Wales Hospital, Shatin, Hong Kong
- National Cancer Center Hospital, Tokyo, Japan
- Singapore (2):
  - National University Hospital Singapore, Singapore
  - National Cancer Centre Singapore, Singapore